CLINICAL TRIAL: NCT00403455
Title: Monoamine Transporters Genotypes: Risk of PTSD and Related Comorbidities
Acronym: MTG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHBA-009-05F; NCT00403455 (Other: Department of Veterans Affairs)
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: PTSD
Keywords: Clinical; Genetics; Monoamine transporter; Pharmacogenetics; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paroxetine Arm (Other): This is a single arm, single site, open-label clinical trial to treat veterans with PTSD. It is a 12-week trial to investigate the efficacy of paroxetine in reducing PTSD symptoms, with the primary outcome measure using CAPS. Genetic information is included to understand why some respond and some do not respond to paroxetine treatment.
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine — SSRI
  Other Names: Paxil

SUMMARY:
Dr. Wang's merit review is aimed at providing a better understanding of the relationship between SLC6A3/SLC6A4 and the mental health of veterans exposed to high levels of combat stress, specifically focusing on PTSD symptoms, related co-morbidities, treatment outcomes and seeks new approaches to therapy for our Veteran population.

DETAILED DESCRIPTION:
Background: Post-traumatic Stress Disorder (PTSD), a debilitating condition that develops following exposure to trauma, is highly prevalent in military personnel and veterans due to high risk of trauma exposure in combat. Trauma exposure, as an environmental insult, is necessary, but itself is not sufficient to cause PTSD, since not everyone exposure to trauma develops PTSD. Brain dopamine (DAT) and serotonin (5-HTT) transporter play a critical role in the regulation of stress related psychological and behavioral functions. Genetic polymorphisms that affect 5-HTT and DAT function, such as the 5' promote polymorphism in the 5-HTT gene (SLC6A4)(5-HTTlpr) and 3' -untranslated region (UTR)-40 bp-variable number tandem repeat (VNTR)of DAT gene (SLC6A3), could influence individual susceptibility to trauma-related psychopathology.

Objective/Hypothesis: The objective of this application is to investigated the relationship between SLC6A3/SLC6A4 and the mental health of veterans exposed to high levels of combat stress, specifically focusing on PTSD symptoms, related comorbidities, and treatment outcome. The central hypothesis is that specific genetic variants that adversely affect serotonin and dopamine neurotransmission constitute a risk for the emergence of PTSD and related comorbid symptoms after trauma exposure; and, some of these variants may further influence PTSD and related response.

Specific Objectives: (1) To determine specific 5-HTTLPR genotype involvement in PTSD symptomatology, (2) to determine influence of combined SLC6A3/SLC6A4 genotypes on PTSD with substance dependence, (3)to identify 5 HTTLPR alleles that affect PTSD symptomatology and treatment outcome, and (4)to identify additional SLC6A3/SLC6A4 alleles associated with PTSD and related comorbidities.

Study Design: We have generated some preliminary data supporting our hypothesis by examining 5-HTTLPR and the 3'-UTR-VNTR of SLC6A3 genotypes in 109 combat veterans with and without PTSD. In this proposal, we will expand on these findings by recruiting 300 veterans exposed to sufficient combat stress defined by Combat Exposure Scale(CES) score of >10 and who qualify for DSM-IV category A PTSD diagnostic criteria, including approximately 150 veterans with PTSD veterans with PTSD defined using DSM-IV diagnostic criteria, Clinician Administered PTSD Scale (CAPS) score >45 and 150 healthy combat-exposed veterans as defined by a CAPS score <15. We will first apply a newly developed extreme discordant phenotype (EDP) method to examine how 5-HTTLPR and 3'-UTR-VNTR genotypes affect trauma related psychopathology in combat veterans only with the highest (>45)and lowest (<15) CAPS scores. Secondly, single nucleotide polymorphisms (SNPs)will be examined across both genes and assessed for relatedness to PTSD susceptibility or resistance. Further analyses of relationship of these polymorphisms with comorbidities will also be performed. Thirdly, a pharmacogenetic trail (using sertraline as a therapeutic agent) will be applied to assess how gene variants influence PTSD treatment outcome. To Safeguard against population stratification, a genome control method will be applied in all the genetic analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female combat veterans ages 18 years and older who meet DSM-III-R criteria for principle diagnosis of PTSD as determined by the CAP-S;
2. A minimum 6-month duration of PTSD illness; 3)CGI-S score of 4 or higher and a total CAPS-2 severity score of 50 or higher at the baseline visit;
3. Homozygous for either the S/S or L/L 5-HTT;
4. Females must not be pregnant or lactating and must agree to an acceptable form of contraception while receiving study medication and for 1 month after.

Exclusion Criteria:

1. Presence of any other primary axis I disorder (concurrent depression will be permitted if it is judged to be secondary to development for PTSD);
2. Suicide ideation or attempts within the past 3 months;
3. Alcohol or substance abuse or dependence in the past six months;
4. Evidence of clinically significant hepatic or renal disease;
5. Previous seizure disorder or condition predisposing to seizures, or on medications that might lower the seizure threshold
6. Any acute or unstable medical condition that might interfere with the safe conduct of the study;
7. Intolerance or hypersensitivity to citalopram or any other SSRI;
8. Treatment with a monoamine oxidase inhibitor within 14 days of initiating the study;
9. Concomitant treatment with serotonin agonists, other SSRIs, meperidine, tramadol or other medication as determined by the study clinician.
10. PTSD symptoms in need of immediate treatment as determined by clinical assessment from a psychiatrist not affiliated with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhewu Wang, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paroxetine Arm: This is a single arm, single site, open-label clinical trial to treat veterans with PTSD. It is a 12-week trial to investigate the efficacy of paroxetine in reducing PTSD symptoms, with the primary outcome measure using CAPS. Genetic information is included to understand why some respond and some do not respond to paroxetine treatment. Both male and female combat veterans ages 18 years and older who meet DSM-III-R criteria for principle diagnosis of PTSD as determined by the CAP-S were recruited for this study.
Period: Overall Study
Arm/Group | Paroxetine Arm
Started | 38
Completed | 37
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The study recruited all veterans that with a CAPS score of >45 and were DSM-IV positive for PTSD. Both males and females with backgrounds in all ethnic groups were aloud to participate in the study.
Arm/Group | Paroxetine Arm
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 48.5789 [25 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: The CAPS assessment is used to determine the severity of an individuals PTSD. The assessment examines Re-experiencing, Avoidance and Numbing, and Hyperarousal symptoms which total score in each of these categories are added together to achieve a total CAPS score. Scores on this assessment can range from 0-136 with 0 not having any PTSD symptoms and 136 having the most symptoms possible. The study uses this assessment at the baseline and at the end of treatment to determine the decrease in this score over the course of the study.
Time Frame: 12 weeks
Population: All participants analyzed had a CAPS score of >45 and were DSM-IV positive for PTSD. Both males and females with backgrounds in all ethnic groups were aloud to participate in the study.
Measure: Mean (Full Range); unit: Change in units on a scale
Arm/Group | Paroxetine Arm
Number analyzed (Participants) | 36
Change in units on a scale | -21.72 [-91 to 30]

ADVERSE EVENTS:
Time Frame: All patients were monitored over a 12 weeks. During this time period no patients experienced any serious adverse events. A small number of participants experienced nausea and other minor symptoms which did not require them stopping the medication.
Description: Paroxetine is and during the time of this study an open-label drug which is approved to treat PTSD. This study was conducted to analyze why some people respond to the medication better than others in relation to a persons genotype.
Arm/Group | Paroxetine Arm
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 11/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paroxetine Arm (N=38)
Minor Nausea (Gastrointestinal disorders) | 11 — All of the non-serious events reported were nausea. All of these patients continued the medication and completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes